CLINICAL TRIAL: NCT01996631
Title: Serum Markers of OS, Inflammation, and EDCs and Impact on the Menstrual Cycle and Reproductive Hormone in Taiwanese Women
Brief Title: The Impact of EDCs Relative Markers and Reproductive Hormone in Taiwanese Women
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Principal Investigator, Ming-I Hsu, Director, Principal Investigator, Taipei Medical University WanFang Hospital
Other Study IDs: Hsu2013-TMU-JIRB 201301040
Record Dates: First submitted 2013-10-21; First posted 2013-11-27 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: Reproductive Aged.

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Oxidative stress(OS), inflammation, and endocrine-disrupting chemicals(EDC) were all thought as important markers that will impact on female reproductive function. However, the cause-result correlations between above parameters were still unclear. Investigator plans to design a study to evaluate the OS, inflammation, and EDC and their impact on the menstrual cycle and reproductive hormone in Taiwanese women. Ferritin is a ubiquitous intracellular protein that is essential for the regulation of iron homeostasis. Serum ferritin level is a widely available clinical biomarker used to estimate body iron status. Iron is a strong pro-oxidant, and high body iron levels are associated with an increased level of OS that may elevate the risk of type 2 diabetes. Mildly elevated body iron stores are associated with statistically significant elevations in glucose homeostasis indexes. Furthermore, patients with elevated iron stores present not only insulin resistance but also metabolic alterations that put them at increased risk of cardiovascular disease. Increased serum ferritin levels have been found in women with Polycystic Ovary Syndrome(PCOS). Serum ferritin were highly correlated with menstrual cycle and androgens level in women. Homocysteine, a sulfur-containing amino acid formed during the metabolism of methionine, exerts cytotoxic effects on the vascular endothelium. Hyperhomocysteinemia has been established as an independent risk factor for thrombosis and cardiovascular disease, and it may partially account for the increased risk of cardiovascular disease associated with insulin resistance. Elevated total plasma homocysteine levels have been established as an independent risk factor for thrombosis and cardiovascular disease. Studies related to homocysteine and PCOS have reported inconsistent results.

Chronic low-grade inflammation has emerged as a key contributor to the pathogenesis of PCOS and obesity. A dietary trigger such as glucose is capable of inciting OS and an inflammatory response from mononuclear cells of women with PCOS, and this phenomenon is independent of obesity. The correlation between inflammatory markers and reproductive endocrine disturbance and consequent complications should be important.Both OS and EDC had been associated with PCOS.

BPA, one of EDC, is an environmental estrogen used in the synthesis of plastics, is a "high-volume production" chemical with widespread human exposure. BPA was been reported in several female reproductive disturbance. However, the pathological pathway of BPA impact on female reproductive system had not been well-understood. Reactive oxygen species have a role in the modulation of gamete quality and gamete interaction. Persistent and elevated generation of ROS leads to a disturbance of redox potential that in turn causes OS. The first part of our study is aim to evaluate the OS impact on the biochemical parameters in women with PCOS; the secondary part of our study is to investigate the BPA on the clinical and biochemical of women with PCOS; finally, investigator plans to test the hypothesis that BPA might increase OS and then elevated ROS in women with menstrual disturbance, furthermore, the role of OS and BPA impact on insulin resistance and metabolic disturbance will be also investigated.

OS, inflammation, and EDCs are all important factors impact on the reproductive competence in women. To clarify above problems are critical importance. Investigator then conduct this study to demonstrate those problems. Study and control cases will be included. Serum total oxidant status, inflammatory biomarkers, total antioxidant status, BPA, and clinical/biochemical parameters will be obtained for all cases. OS and BPA will be evaluated with all clinical/biochemical parameters for all subjects.

ELIGIBILITY:
Inclusion Criteria:

* Reproductive aged women.

Exclusion Criteria:

* Clinical diagnosed of congenital adrenal hyperplasia, androgen-secreting tumor, Cushing's syndrome, Asherman's syndrome, Mullerian agenesis, and chromosomal anomalies;
* Menarche in 1 years and older than 49;
* Hormones or drugs for major medical diseases used.

Ages: 20 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients who are reproductive aged and come visit our OPD clinic, except postmenopausal and before menarche.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2013-06; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Endocrine-disrupting chemicals | The study will start from June 6, 2013 to May 31, 2016, up to 3 years.
  To study the correlation between serum markers of oxidative stress, inflammation, and endocrine-disrupting chemicals (EDCs) and their impact on the menstrual cycle and reproductive hormone in Taiwanese women.

CONTACTS AND LOCATIONS:
Overall Officials: Ming I Hsu, MD, Principal Investigator — Taipei Medical University WanFang Hospital